CLINICAL TRIAL: NCT03336164
Title: Impact of a Front-of-pack Nutrition Label on the Nutritional Quality of Purchases in Campus University Restaurant
Brief Title: FOP Nutrition Label in Campus Campus University Restaurant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Responsible Party: Principal Investigator, Mathilde Touvier, Head of Department, University of Paris 13
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CROUS_NICE2R
Record Dates: First submitted 2017-11-03; First posted 2017-11-08 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Food Labelling

STUDY DESIGN:
Intervention Model Description: After a control period with no specific front-of-pack labeling, the intervention consists in the apposition of a front-of-pack labeling (Nutri-Score) to individual foods in a campus university restaurant. All foods are individually labeled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Front-of-pack labelling Nutri-Score (Experimental): Introduction of the Nutri-Score front-of-pack nutrition label on every food and beverage sold in the same campus university restaurant after the control period without food labelling.
  The implementation of the label is accompanied by a communication campaign towards students in the form of posters and leaflets.
  Interventions: Behavioral: Front-of-pack labelling Nutri-Score

INTERVENTIONS:
Behavioral: Front-of-pack labelling Nutri-Score — Introduction of the Nutri-Score front-of-pack nutrition label on shelf display tags for every food and beverage sold in the university restaurant

SUMMARY:
This study evaluates the impact of the introduction of a front-of-pack nutrition label on foods and beverages sold in a campus university restaurant in France on the nutritional quality of purchases.

DETAILED DESCRIPTION:
The introduction of front-of-pack nutrition labelling is thought to help consumers making healthier food choices at the point-of-purchase.

Recently, the French government has selected the Nutri-Score as single front-of-pack nutrition label.

Evaluations of the Nutri-Score suggest it is helping consumers making healthier choices. However, its impact in vulnerable populations has not yet been tested. Students are thought to be a vulnerable population due to their limited resources and to their unhealthy food choices.

The objective of the present study is to investigate the impact of the introduction of the Nutri-Score in campus university restaurant on the nutritional quality of food purchases. The intervention is conducted during several months, with a control period without front-of-pack nutrition labelling at the beginning of the university year.

Data on purchases is collected regularly through receipts, and the nutritional quality of purchases is evaluated over time between the intervention situation and the control situation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects purchasing foods or beverages in the selected campus university restaurant

Exclusion Criteria:

* None No individual data is collected. Only purchases data is collected (cash register sales data)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-05-27 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Overall nutritional quality of purchases | Every 15 days, up to 6 months
  Overall nutritional quality of purchases evaluated using the Food Standard Agency nutrient profiling system

SECONDARY OUTCOMES:
Energy content of purchases | Every 15 days, up to 6 months
  Energy content of the purchases (kcal/100g)
Saturated fat content of purchases | Every 15 days, up to 6 months
  Saturated fat content of the purchases (g/100g)
Sugar content of purchases | Every 15 days, up to 6 months
  Sugar content of the purchases (g/100g)
Sodium content of purchases | Every 15 days, up to 6 months
  Sodium content of the purchases (g/100g)
Fiber content of purchases | Every 15 days, up to 6 months
  Fiber content of the purchases (g/100g)
Protein content of purchases | Every 15 days, up to 6 months
  Protein content of the purchases (g/100g)

CONTACTS AND LOCATIONS:
Locations (1):
- CROUS Nice - Toulon, Nice, France

IPD SHARING:
Plan to Share IPD: No